CLINICAL TRIAL: NCT00342966
Title: Characterization of the Pharmacokinetics of Oral Selenium Compounds in Humans Before and Following Supplementation
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999999032; OH99-C-N032
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-07-23

CONDITIONS: Cancer
Keywords: Metabolism; Tracer Studies; Chemoprevention; Selenomethionine; Plasma Selenoproteins
MeSH Terms: conditions — Neoplasms

SUMMARY:
The chemopreventive efficacy of Se was tested in a 10-year human intervention trial; total and lung cancer mortality, total cancer incidence, colorectal cancer and prostate cancer incidence decreased. This study is designed to compare, via stable isotope tracer studies the kinetics of inorganic and organic Se before and following two years of oral supplementation with L-selenomethionine, to measure forms of Se in the plasma (extracellular Se-dependent glutathione peroxidase [GSHPx], selenoprotein-P [SeP], albumin-bound Se [AlbSe] and nonprotein-bound low molecular weight [LMWSe] fractions), and to determine the effects of supplementation on the ecology of the hindgut microflora. The forms of Se were chosen to resemble the metabolism of the principal forms of Se in mixed American diets. Sodium selenite, an inorganic form, is metabolized by reduction to selenide which is then either used in the co-translational synthesis of SeCys in specific Se-containing proteins (e.g., glutathione peroxidases, diodinases, selenoproteins P and W), or is converted to methylated excretion products; in this sense it resembles the food form selenocysteine (SeCys) which is metabolized to the selenide level. Selenomethionine (SeMet), an organic form, is a major form of Se in many foods, particularly those of plan origin. In addition to being metabolized to selenide, SeMet also enters the metabolic protein pool by competing with the sulfur-containing amino acid, methionine. A study is proposed to assess the impact of selenium (Se) supplementation on its metabolism in humans.

A pilot study will be conducted to test recruitment strategies and sample collection, preparation and analysis and to assess the detectability of two stable isotopes given together. Four subjects will receive two 300 ug oral doses consisting of 150 ug of the stable isotope 76Se as selenite and 150 ug of the stable isotope 74Se as selenomethionine on study days one and twelve. Subjects will be followed for six weeks.

In the first pharmacokinetics tracer study (PK1), twenty-eight subjects will receive the same two labeled stable isotope doses, and will be followed for 4 months. In addition, two subjects who have been self-supplementing with 200 ug of Se as selenized yeast for two years will take part in PK1 to assess the sensitivity over time of the tracer assay in supplemented subjects. PK1 will be followed by a 2-yr supplementation period, in which all 28 subjects will receive daily doses of 200 ug of L0SeMet; subjects = metabolism is expected to approach a new steady state reflective of long-term supplementation. A second 4-month pharmacokinetic tracer study (PK2) will then be conducted while subjects remain on Se-supplementation with an extension of six monthly blood samples. Extensive sampling of plasma, urine, and feces during PK1 and PK2 will permit both the refinement of existing baseline models for selenite and selenomethionine metabolism in humans and the investigation of changes in metabolism arising from Se-supplementation. The study is designed to detect a difference of 0.75 standard deviation units in pre-versus post-supplementation rate parameters, assuming a two-sided test with an alpha level of 0.05 and a power of 0.80.

The non-absorbed portion of Se may favor portions of the normal colonic bacterial microflora that produce certain short-chain fatty acids that colon cells use for energy. To test this hypothesis, fecal specimens will be analyzed for short-chain fatty acids over the course of Se-supplementation. In addition, the sampling of buccal cell-Se and of toenail-Se on a quarterly basis over the course of the study and assay of thyroid hormone levels during the first year of the study will permit the investigation of possible changes in levels resulting from supplementation.

DETAILED DESCRIPTION:
The chemopreventive efficacy of Se was tested in a 10-year human intervention trial; total and lung cancer mortality, total cancer incidence, colorectal cancer and prostate cancer incidence decreased. This study is designed to compare, via stable isotope tracer studies the kinetics of inorganic and organic Se before and following two years of oral supplementation with L-selenomethionine, to measure forms of Se in the plasma (extracellular Se-dependent glutathione peroxidase [GSHPx], selenoprotein-P [SeP], albumin-bound Se [AlbSe] and nonprotein-bound low molecular weight [LMWSe] fractions), and to determine the effects of supplementation on the ecology of the hindgut microflora. The forms of Se were chosen to resemble the metabolism of the principal forms of Se in mixed American diets. Sodium selenite, an inorganic form, is metabolized by reduction to selenide which is then either used in the co-translational synthesis of SeCys in specific Se-containing proteins (e.g., glutathione peroxidases, diodinases, selenoproteins P and W), or is converted to methylated excretion products; in this sense it resembles the food form selenocysteine (SeCys) which is metabolized to the selenide level. Selenomethionine (SeMet), an organic form, is a major form of Se in many foods, particularly those of plan origin. In addition to being metabolized to selenide, SeMet also enters the metabolic protein pool by competing with the sulfur-containing amino acid, methionine. A study is proposed to assess the impact of selenium (Se) supplementation on its metabolism in humans.

A pilot study will be conducted to test recruitment strategies and sample collection, preparation and analysis and to assess the detectability of two stable isotopes given together. Four subjects will receive two 300 ug oral doses consisting of 150 ug of the stable isotope 76Se as selenite and 150 ug of the stable isotope 74Se as selenomethionine on study days one and twelve. Subjects will be followed for six weeks.

In the first pharmacokinetics tracer study (PK1), twenty-eight subjects will receive the same two labeled stable isotope doses, and will be followed for 4 months. In addition, two subjects who have been self-supplementing with 200 ug of Se as selenized yeast for two years will take part in PK1 to assess the sensitivity over time of the tracer assay in supplemented subjects. PK1 will be followed by a 2-yr supplementation period, in which all 28 subjects will receive daily doses of 200 ug of L0SeMet; subjects = metabolism is expected to approach a new steady state reflective of long-term supplementation. A second 4-month pharmacokinetic tracer study (PK2) will then be conducted while subjects remain on Se-supplementation with an extension of six monthly blood samples. Extensive sampling of plasma, urine, and feces during PK1 and PK2 will permit both the refinement of existing baseline models for selenite and selenomethionine metabolism in humans and the investigation of changes in metabolism arising from Se-supplementation. The study is designed to detect a difference of 0.75 standard deviation units in pre-versus post-supplementation rate parameters, assuming a two-sided test with an alpha level of 0.05 and a power of 0.80.

The non-absorbed portion of Se may favor portions of the normal colonic bacterial microflora that produce certain short-chain fatty acids that colon cells use for energy. To test this hypothesis, fecal specimens will be analyzed for short-chain fatty acids over the course of Se-supplementation. In addition, the sampling of buccal cell-Se and of toenail-Se on a quarterly basis over the course of the study and assay of thyroid hormone levels during the first year of the study will permit the investigation of possible changes in levels resulting from supplementation.

ELIGIBILITY:
* INCLUSION CRITERIA:

Those subjects with normal physical examinations and Se plasma levels within the eligible range will be invited to participate in the study.

Men and women will be recruited according to the following eligibility criteria. Subjects must:

be between the ages of 20 and 60 years;

be in general good health as determined by a screening history and physical examination and laboratory tests with no history of gastrointestinal, hepatic, renal and/or hematologic diseases, cancer, coronary heart disease;

be within 20% from their ideal weight as described in the Metlife Height and Weight Tables (1993);

be consuming typical mixed diets;

give informed consent; and

be judged, based on a personal interview, as having a high probability of participating for the two-year eight month duration of the study.

EXCLUSION CRITERIA:

women: pregnant or lactating women; sexually active and not using contraceptives (e.g., condoms, oral contraceptives, diaphragm); planning to become pregnant during the experimental period; or post -menopausal (at least 6 months);

taking antibiotics on a regular basis;

have a history of taking Se supplements of more than 25 ug/d in the past year;

current smoker, or stopped smoking within the last 6 months;

on rigorous exercise or weight-reduction programs.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 1999-06-14; Study Completion 2010-07-23

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - USDA, Beltsville, Maryland
  - National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Ankerst J, Sjogren HO. Effect of selenium on the induction of breast fibroadenomas by adenovirus type 9 and 1,2-dimethylhydrazine-induced bowel carcinogenesis in rats. Int J Cancer. 1982 Jun 15;29(6):707-10. doi: 10.1002/ijc.2910290618. PMID 7107071
- [Background] Bergad PL, Rathbun WB. Inhibition of Na,K-ATPase by sodium selenite and reversal by glutathione. Curr Eye Res. 1986 Dec;5(12):919-23. doi: 10.3109/02713688608995172. PMID 3026732
- [Background] Birt DF, Julius AD, Runice CE, White LT, Lawson T, Pour PM. Enhancement of BOP-induced pancreatic carcinogenesis in selenium-fed Syrian golden hamsters under specific dietary conditions. Nutr Cancer. 1988;11(1):21-33. doi: 10.1080/01635588809513966. PMID 2832833